CLINICAL TRIAL: NCT06330948
Title: Effects of SugarCut® Unripe Guava Fruit Extract on Blood Glucose Regulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, YenPing, Lei, Assistant professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NYCU112183AEF
Record Dates: First submitted 2024-03-05; First posted 2024-03-26 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo group (Placebo Comparator): Placebo group (50mL/bottle)
  Interventions: Dietary Supplement: Placebo group
- SugarCut® Unripe Guava Fruit Extract (Experimental): SugarCut® Guava Fruit Extract Group (50mL/bottle, each bottle contains 10g Guava Fruit Extract)
  Interventions: Dietary Supplement: SugarCut® Unripe Guava Fruit Extract

INTERVENTIONS:
Dietary Supplement: SugarCut® Unripe Guava Fruit Extract — This trial adopted a double-blind placebo-controlled parallel testing design. Subjects will be randomly assigned to the SugarCut® Guava Extract group. Before the trial (week 0), subjects are required to undergo fasting blood collection and height, weight, and blood pressure examinations. Afterwards, the test samples were given to the subjects for 8 consecutive weeks, and they were reviewed for evaluation at the 4th and 8th weeks, and fasting blood collection and height, weight, and blood pressure examinations were performed.
  Arms: SugarCut® Unripe Guava Fruit Extract
Dietary Supplement: Placebo group — This trial adopted a double-blind placebo-controlled parallel testing design. Subjects will be randomly assigned to the placebo group. Before the trial (week 0), subjects are required to undergo fasting blood collection and height, weight, and blood pressure examinations. Afterwards, the test samples were given to the subjects for 8 consecutive weeks, and they were reviewed for evaluation at the 4th and 8th weeks, and fasting blood collection and height, weight, and blood pressure examinations were performed.
  Arms: placebo group

SUMMARY:
Guava (Psidium guajava) belongs to the Myrtle family. It is a tropical and subtropical fruit native to the Americas. Ripe guava fruit is sweet and delicious. It is rich in vitamins A, C and trace elements such as phosphorus, calcium and magnesium. In traditional medicine, guava fruit can be eaten raw, and the roots can treat stomach problems, abdominal pain, dysentery, and diabetes; the leaves can treat diabetes, abdominal pain, rheumatism, antipyretic, stomachache, anthelmintic, cholera, vomiting, diarrhea, enteritis and other symptoms. Guava leaf extract contains polyphenols. Studies have shown that guava leaf has antioxidant, blood sugar regulating and anti-cancer effects. Not only guava leaves, research has found that guava fruits are rich in vitamins, fiber and antioxidants, which have anti-inflammatory and anti-cancer effects. Preliminary research has found that the extract of red guava young fruit has more active ingredients - saponins and total polyphenol content, and its antioxidant capacity is also higher than that of mature guava. In vitro studies have found that guava fruit extract can increase the expression of GLUT4 gene and promote the entry of blood sugar into cells. At the same time, guava fruit extract can inhibit the formation of final glycated proteins (AGEs). The purpose of this study is to explore the effect of guava fruit extract on blood sugar regulation in humans and to evaluate its potential to be developed as a blood sugar regulation supplement.

DETAILED DESCRIPTION:
This trial adopted a double-blind placebo-controlled parallel testing design. Subjects will be randomly assigned to the placebo group and the SugarCut® Guava Extract group, with 30 people in each group. Before the trial (week 0), subjects are required to undergo fasting blood collection and height, weight, and blood pressure examinations. Afterwards, the test samples were given to the subjects for 8 consecutive weeks, and they were reviewed for evaluation at the 4th and 8th weeks, and fasting blood collection and height, weight, and blood pressure examinations were performed.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 20-60.
2. Fasting blood glucose level is between 100 ~ 126 mg/dL.

Exclusion Criteria:

1. Patients with renal insufficiency and kidney dialysis.
2. Cancer patients.
3. Those taking blood sugar regulation-related drugs.
4. Have a history of guava allergy
5. People suffering from mental illness
6. Pregnant and breastfeeding women
7. Long-term use of blood sugar regulating supplements

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
GLUT4 gene expression | Week 4 and 8
  GLUT4 expression is exquisitely regulated in muscle and this seems important in the regulation of insulin-stimulated glucose uptake by this tissues. Thus, muscle GLUT4 overexpression in transgenic animals ameliorates insulin resistance associated with obesity or diabetes.
Hematology Test | Week 4 and 8
  Fasting blood glucose, HbA1c, insulin, final glycated proteins (AGEs), triglycerides, total cholesterol, Blood urea nitrogen, Creatinine, Uric acid, GOT, GPT, Low glucagon-like peptide-1 (GLP-1)

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Beitou Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No